CLINICAL TRIAL: NCT00051545
Title: Seocalcitol Versus Placebo in the Adjuvant Treatment of Hepatocellular Carcinoma. Efficacy of Seocalcitol (EB 1089) Enteric-Coated Capsules (5 ug) or Placebo in Prolonging Time to Relapse Following Intended Curative Resection or Percutaneous Ablative Treatment for Hepatocellular Carcinoma
Brief Title: Seocalcitol Versus Placebo in the Adjuvant Treatment of Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EBC 9802 INT
Record Dates: First submitted 2003-01-13; First posted 2003-01-14 (Estimated); Last update posted 2025-02-25 (Actual); Status verified 2005-04

CONDITIONS: Liver Neoplasms
Keywords: liver; cancer; hepatocellular; carcinoma
MeSH Terms: conditions — Liver Neoplasms; Neoplasms; Carcinoma | interventions — seocalcitol

INTERVENTIONS:
Drug: Seocalcitol

SUMMARY:
To evaluate the efficacy of Seocalcitol in prolonging time to relapse following intended curative resection or percutaneous ablative treatment, i.e. percutaneous ethanol injection(s), percutaneous acetic acid injection(s), percutaneous microwave coagulation therapy, or percutaneous radiofrequency ablation for hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* Hospital in- or out patients
* Either sex
* 18 to 75 years of age
* With hepatocellular carcinoma treated successfully with surgical resection or percutaneous ablative treatment within 4 and 8 weeks, respectively, prior to inclusion.
* All patients must give their signed informed consent to join the study.

Exclusion Criteria:

* Patients previously treated with any anti-cancer therapy for HCC except for surgical resection and percutaneous ablative therapy
* Patients treated with chemotherapy or other anti-cancer therapy (except surgical resection or percutaneous ablative treatment) in the previous 4 weeks
* Patients with another primary tumor except basocellular carcinoma of the skin or in situ carcinoma of the cervix within the last 2 years
* With a history of renal stone(s)
* With a life expectancy < 3 months
* WHO performance status 3 or 4.
* Patients with hypercalcemia (ionised serum calcium > 1.35 mmol/l or albumin corrected serum calcium > 2.68 mmol/l), previous/current calcium metabolic disease, taking calcium-lowering therapy or medication known to affect systemic calcium metabolism, or with marked laboratory abnormalities.
* Patients with recurrent hepatocellular carcinoma, with known extrahepatic metastases, Okuda stage III disease and patients with a Child-Pugh score of C are also excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608
Dates: Start 1999-11; Study Completion 2004-06

PRIMARY OUTCOMES:
Time to relapse, relapse being defined as the first recurrence of HCC (intra- or extrahepatic).

SECONDARY OUTCOMES:
Survival
Time to distant recurrence of HCC
Time to second primary HCC
Time to development of metastases
Tumour measurements
Tumour marker (alpha-fetoprotein AFP)
Quality of life
Length of hospital stay
Adverse events
Laboratory safety examinations
Dose of Seocalcitol

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Hvidberg, MScPharm PhD, Study Director — LEO Pharma
Locations (5):
- E.g., University Health Network Toronto General Hospital (numerous facilities in Canada are recruiting), Toronto, Ontario, Canada
- E.g., Hopital Notre-Dame de Bon Secour, Service de Hepato-gastro-enterologie (numerous facilities are recruiting in France), Metz, France
- E.g., Osp. Maggiore, Policlinico di Milano, Divisione di Medicina Interna (numerous facilities are recruiting in Italy), Milan, Italy
- E.g. Hospital Clinic Provincial de Barcelona (numerous facilities are recruiting in Spain), Barcelona, Spain
- E.g., The University of Edinburgh Royal Infirmary (numerous facilities are recruiting in UK), Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en